## Public messaging to increase treatment seeking among Veterans at risk for suicide during transition from military service

NCT04784663

July 17, 2025

**Overview:** This is a national VA research study conducted by the Center of Excellence at the VA Finger Lakes Healthcare System in New York. The purpose of the study to better understand how to reach and engage Veterans who recently discharged from the U.S. military with suicide prevention campaigns to encourage help seeking. To do so, we are asking Veterans across the country their opinions and beliefs on what types of public messages they think work and don't work. Your responses will help us to learn more about VA campaigns and potentially improve these types of initiatives to better meet the needs of new Veterans. This study is approved by the IRB (research review committee) (Study ID # 1551390) and is funded by a research grant awarded from VA Health Services Research & Development (Grant # SDR-19-354).

You were invited to take part in this research because you served in the U.S. military and discharged in the past year. We estimate that up to 600 Veterans across the U.S. will take part in this study. All study procedures occur virtually at your convenience – you are not expected to visit a VA Medical Center for any tasks and will work with you to complete the study at a time that works for you. This research project is independent of any health care or benefits at the VA.

**Study Description:** You will need to download and use the study's free mobile app on your own reliable Smartphone to participate. If you decide to take part in this study, you will spend approximately 1-1.5 hours each month completing study tasks for the next 2 months from beginning to end. Your involvement begins with our telephone survey today that will take about an hour. This survey will ask you what you think about VA suicide prevention messaging, your awareness of VA campaigns as well as attitudes and behaviors related to mental health and help seeking. No identifiable or personal health information is collected as part of this survey. You will complete similar surveys by telephone two more times with research staff, approximately 1 and 2-months from now. You may also be asked several additional open-ended questions during your 2-month survey related to your experience in the study including the use of the study's Smartphone app. We will contact you several weeks ahead of time to schedule at a time convenient to you.

I will then randomly assign you to 1 of our 3 study groups. These groups participate in different ways to help our researchers examine our suicide prevention messages. Then we will download the study mobile app together to your phone from your App Store, and I will give you a code to 'activate' the app on your phone. We will then go through how to use the app, and I can answer any questions you might have. I will also provide you with information on how to service the mobile app if it malfunctions during your participation. It is important that you know the mobile app requires internet access (WiFi) or cellular data connection to function. Of note, the VA will not reimburse you for any of charges related to mobile phone or internet access.

The mobile app will send you weekly push notifications. At some point during the 2-month study period, you will also receive 4 short study videos, each less than 2 minutes long, to watch through the mobile app as well. When you receive these videos will be dependent on the group you were assigned to by me.

**Compensation:** You will be compensated up to \$75 for your time completing the surveys and watching video messages by VA check or direct deposit. Funds are distributed following each assessment: \$20 at baseline (today), \$25 following the 1-month telephone survey, and \$30 following the 2-month telephone survey. I will collect information required to process payment at the end of our call today. You will receive payments within 6-10 weeks of voucher processing. It is important for you to know that payments for participation in a study are taxable income. There is not cost associated with participation in this study. If you voluntarily end participation early or

the research staff makes the determination that your participation in the study is causing you harm, you will be paid for your time for the study activities you completed.

**Participation Risks/Benefits:** Research participation could have some possible risks or discomforts. While no physical risks are expected as part of participation in this study, you will be asked to answer questions that could upset you such as items related to your health, attitudes, behaviors and how you handle stress. There is the possibility that the study messages could make you feel uncomfortable. If you experience distress at any time, the research team can work with you to make you feel more comfortable. You may also skip any questions you don't want to answer. If you continue to feel distressed, researchers may end your participation. There is the potential risk for loss of confidentiality or privacy. However, a random subject number will be assigned to your responses to enhance confidentiality of your answers.

Identifiable information (i.e., your name, payment information, etc.) and data are never linked for research purposes and are stored separately to enhance confidentiality. If results of the study are reported in research journals or at research meetings, you will not be identified by name or any other means but rather data is reported in aggregate form (all responses from participants are combined together). The data you provide could be used by another researcher for future research studies without your or your legally authorized representative's consent. Should this happen, information that could personally identify you will be removed. In fact, other researchers are prohibited from identifying any individuals in the study.

There is no guarantee of direct benefit to you by participating as this study is not designed to treat illness or to improve your health. But your responses may help other Veterans by informing the design of future VA suicide prevention campaigns and outreach.

**Safety Protocol:** If there is any indication of risk for suicide or violence or other threats to safety, then the research team may break confidentiality and take actions to promote safety. These actions may include consulting with the police or emergency services or connecting you to the Veterans Crisis Line for further assessment and potential emergency intervention. At any time, you may also contact the Veterans Crisis Line by phone (call 988 and press 1), or your own doctor to alleviate concerns. If you are ever at immediate risk or harm, please call 9-1-1.

**Voluntary Nature:** Participation in this study is completely voluntary, and your decision to participate will have no impact on VA healthcare, services, or benefits. You are free to withdraw at any time during the study. You can call the study's toll-free number at --- and leave a message with your name and phone number to let us know you no longer would like to participate.

**Data Security:** Only approved research team members with a 'need to know' will have access to any study data. Any paper records are kept in a secure facility in locked filing cabinet in locked offices in the Center of Excellence within the VA Finger Lakes Healthcare System in NY. Any electronic information collected is kept on secure password-protected VA computers on servers behind VA computer security systems (firewall).

The company that has developed the study's Smartphone App cannot identify you personally, will have none of your information, and are not permitted to use or sell data.

**Study Contacts**: If you have any questions or concerns about this study you can reach the research team toll free at any time at ---. This number was also provided on the invitational letter

you received for this study. Also, you can reach the Chair of the VA Institutional Review Board (IRB). An IRB is a group of people who perform independent review of research studies.

You might want to contact the IRB about such issues as:

- You have questions, concerns, or complaints that are not being answered by the research team
- You are not getting answers from the research team
- You cannot reach the research team
- You want to talk to someone else about the research
- You have questions about your rights as a research participant